CLINICAL TRIAL: NCT03765138
Title: Combined Prolonged Exposure and Pramipexole Treatment for Patients With PTSD and Depression
Brief Title: Combined Treatment of Prolonged Exposure and Pramipexole for Posttraumatic Stress Disorder and Depression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Patient recruitment difficulties
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor of Medical Psychology, Research Foundation for Mental Hygiene, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Research Foundation for Mental
Record Dates: First submitted 2018-12-02; First posted 2018-12-05 (Actual); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: PTSD; MDD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PE/Pramipexole (Experimental): Experimental: Prolonged Exposure/Pramipexole Prolonged Exposure (PE) Therapy consists of 10 sessions of 90-minute duration, normally conducted once a week. In addition to receiving PE as described above, patients will have Pramipexole treatment.
  Interventions: Combination Product: PE/Pramipexole

INTERVENTIONS:
Combination Product: PE/Pramipexole — Experimental: PE/Pramipexole Prolonged Exposure (PE) Therapy consists of 10 sessions of 90-minute duration, normally conducted once a week. Elements of PE include imaginal and in vivo exposure to trauma reminders; breathing retraining; cognitive restructuring; and PTSD psychoeducation.
  Pramipexole: In addition to receiving PE as described above, patients will have Pramipexole treatment. Daily dose will be started at 0.25 mg/day and increased by 0.25 mg/day every 3-4 days to a target of 2.5mg day by week 5. Beginning week 6 daily dose will be increased weekly by 0.5 mg/day to a maximum dose of 4mg. Dose will be increased as tolerated unless the patient has achieved remission and will be decreased in the event of intolerable adverse events.

SUMMARY:
This pilot study aims to test the safety, feasibility, and initial efficacy of combined 10 week treatment of prolonged exposure (PE) and Pramipexole in patients with comorbid posttraumatic stress disorder (PTSD) and depression (MDD). Resting state functional connectivity (rsFC) will be assessed at baseline and en of treatment.

DETAILED DESCRIPTION:
Approximately half of the individuals with posttraumatic stress disorder (PTSD) present with major depressive disorder (MDD). Compared to PTSD alone, patients with comorbid PTSD-MDD demonstrate greater distress and poorer treatment outcome. Functional magnetic resonance imaging (fMRI) show that relative to PTSD alone, PTSD-MDD is associated with decreased resting state functional connectivity (rs-FC) in both fear- and reward-processing circuits. In addition, our data suggest that Prolonged Exposure (PE), first-line PTSD treatment, may successfully target impairments in the fear circuits, but not in the reward circuits, which may explain the treatment-refractory quality of PTSD-MDD.

The goal of this pilot study is to test the feasibility, safety and initial efficacy of an integrated therapeutic approach targeting both fear and reward impairments in PTSD-MDD patients. Specifically, the investigators will examine a combination treatment with PE, shown to effectively address fear circuitry deficits, and Pramipexole, a dopamine agonist, shown to increase reward circuit function and to have promise in treating depression but not previously studied in PTSD. The central hypothesis is that combined PE/Pramipexole will a) improve PTSD and depressive symptoms in PTSD-MDD patients, and b) increase functional connectivity of fear and reward pathways as measured by fMRI rs-FC. In this pilot study, 15 adults aged 18-60 years with PTSD-MDD will receive combined 10-week of PE and Pramipexole up to the maximum dose of 4mg a day. Clinical assessment will be conducted at baseline, week 5, post treatment and at 3-month follow up. Behaviorally assessments including the probabilistic reward task (PRT) and attention allocation tasks, and fMRI scans for resting state functional connectivity (rs-FC) will be conducted at baseline and end of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 60
2. Current DSM-V diagnosis of PTSD comorbid with MDD
3. CAPS-5 ≥ 25, and 17-item HRSD ≥ 17
4. Able to give consent, fluent in English

Exclusion Criteria:

1. Prior or current diagnosis with traumatic brain injury, bipolar disorder, psychotic disorder, gambling or impulse control disorders, or dementia
2. History of psychosis, psychotic disorder, mania or bipolar disorder
3. Severe substance use disorder excluding nicotine (i.e., nicotine use disorder and mild-moderate alcohol/cannabis use disorder are accepted)
4. Individuals at risk for suicide based on history and current mental state. BDI-II suicide item > 2 or CGI-Severity baseline score of 7.
5. Treatment with antidepressants or other psychotropic medication in the past 4 weeks (or 6 weeks for fluoxetine; an exception will be made for zolpidem used intermittently for sleep).
6. Pregnancy or plans to become pregnant during the period of the study.
7. Current psychotherapy
8. Current unstable or untreated medical illness
9. Any condition that would exclude clinical MRI exam (e.g. pacemaker, paramagnetic metallic prosthesis, surgical clips, shrapnel, necessity for constant medicinal patch, some tattoos, severe obesity, claustrophobia)
10. History of untoward reaction to pramipexole

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — Columbia Psyhciatry and New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: PTSD Research and Treatment Program at Columbia Psychaitry — https://www.columbiapsychiatry.org/research-clinics/ptsd-research-and-treatment-program

RESULTS

PARTICIPANT FLOW:
Groups:
- PE/Pramipexole: Experimental: Prolonged Exposure (PE)/Pramipexole PE Therapy consists of 10 sessions of 90-minute duration, normally conducted once a week. In addition to receiving PE as described above, patients will have Pramipexole treatment.
  PE/Pramipexole: Experimental: PE/Pramipexole PE Therapy consists of 10 sessions of 90-minute duration, normally conducted once a week. Elements of PE include imaginal and in vivo exposure to trauma reminders; breathing retraining; cognitive restructuring; and PTSD psychoeducation.
  Pramipexole: In addition to receiving PE as described above, patients will have Pramipexole treatment. Daily dose will be started at 0.25 mg/day and increased by 0.25 mg/day every 3-4 days to a target of 2.5mg day by week 5. Beginning week 6 daily dose will be increased weekly by 0.5 mg/day to a maximum dose of 4mg. Dose will be increased as tolerated unless the patient has achieved remission and will be decreased in the event of intolerance.
Period: Overall Study
Arm/Group | PE/Pramipexole
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | PE/Pramipexole
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms as Measured by the Clinician Administered PTSD Scale for DSM-5 (CAPS-5)
Description: The CAPS is the gold standard in PTSD assessment. It is a 30-item structured interview used for current (past week or month) and lifetime diagnosis of PTSD. The CAPS was designed to be administered by clinicians and clinical researchers who have a working knowledge of PTSD. The full interview takes 45-60 minutes to administer. Scores range from 0 to 80 with higher values represent a worse outcome.
Time Frame: Baseline, Week 5, Week 10, 3 month follow up
Population: Participant did not complete protocol.
Arm/Group | PE/Pramipexole
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Depressive Symptoms as Measured by the Hamilton Rating Scale for Depression (HRSD).
Description: The Hamilton Rating Scale for Depression is a 17-item instrument that was designed to measure frequency and intensity of depressive symptoms in individuals with major depressive disorder. Ratings are made using either a five- or a three-point scale, yielding total scores from 0 to 61, with higher values represent a worse outcome.
Time Frame: Baseline, Week 5, Week 10, 3 month follow up
Population: Study discontinued
Groups:
- PE/Pramipexole: Experimental: Prolonged Exposure/Pramipexole Prolonged Exposure (PE) Therapy consists of 10 sessions of 90-minute duration, normally conducted once a week. In addition to receiving PE as described above, patients will have Pramipexole treatment.
  PE/Pramipexole: Experimental: PE/Pramipexole Prolonged Exposure (PE) Therapy consists of 10 sessions of 90-minute duration, normally conducted once a week. Elements of PE include imaginal and in vivo exposure to trauma reminders; breathing retraining; cognitive restructuring; and PTSD psychoeducation.
  Pramipexole: In addition to receiving PE as described above, patients will have Pramipexole treatment. Daily dose will be started at 0.25 mg/day and increased by 0.25 mg/day every 3-4 days to a target of 2.5mg day by week 5. Beginning week 6 daily dose will be increased weekly by 0.5 mg/day to a maximum dose of 4mg. Dose will be increased as tolerated unless the patient has achieved remission.
Arm/Group | PE/Pramipexole
Number analyzed (Participants) | 0

3. Secondary Outcome: Changes in Functional Connectivity of Fear and Reward Pathways as Measured by Functional Magentic Resonance Imaging (fMRI) Resting State Functional Connectivity (Rs-FC).
Description: The investigators will use fMRI scans at baseline and posttreatment to assess connectivity in fear and reward circuits
Time Frame: baseline and week 10.
Population: Study discontinued
Arm/Group | PE/Pramipexole
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 5 months
Arm/Group | PE/Pramipexole
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT03765138/Prot_SAP_000.pdf